CLINICAL TRIAL: NCT03520114
Title: Randomized Trial of Retropubic Versus Single-incision Mid-Urethral Sling (Altis ) for Concomitant Management of Stress Urinary Incontinence During Native Tissue Vaginal Repair
Brief Title: Retropubic vs. Single-Incision Mid-Urethral Sling for Stress Urinary Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Foundation for Female Health Awareness (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00050256
Record Dates: First submitted 2018-04-26; First posted 2018-05-09 (Actual); Results first posted 2025-01-16 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2023-09

CONDITIONS: Stress Urinary Incontinence; Pelvic Floor Disorders
Keywords: Retropubic sling; Single-incision sling; Vaginal repair; Management
MeSH Terms: conditions — Urinary Incontinence, Stress; Pelvic Floor Disorders

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants and will be masked during the one-year follow-up period.Precautions will be taken to minimize unmasking the study groups: Since RP slings require two suprapubic stab incisions, identical sham incision will also be performed in the SIS group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- RP sling group (Experimental): Participants assigned to the retropubic (RP) sling group will have the RP sling placement procedure.
  Interventions: Device: RP sling placement
- SIS group (Experimental): Participants assigned to the single-incision sling (SIS) group will have the SIS placement procedure.
  Interventions: Device: SIS placement

INTERVENTIONS:
Device: RP sling placement — A 1.5 cm incision will be made at the mid-urethra through a separate vaginal incision with lateral dissection with Metzembaum scissors. After placement of both trocars, cystoscopy with a 70-degree scope will be performed to assess for bladder and urethral injury. Surgeons will set the tension of the tension-free vaginal tape (TVT) slings so that a spacer can be placed between the sling and the urethra. Sling tensioning will be performed after anterior and apical prolapse is corrected.
  Arms: RP sling group
Device: SIS placement — The sling is introduced through a single anterior vaginal incision of 1.5 cm at the mid-urethra. The sling/needle assembly is advanced behind the ischiopubic rami in a transobturator trajectory toward the obturator space bilaterally. The needle is then removed by simply sliding the fixating tip back out. The other side is then completed in an identical fashion. After the fixation of the two anchors at the 2 and 10 o'clock positions, the patient's bladder is filled with 250 mL of Sodium Chloride (NaCl). Afterward, an intraoperative crede maneuver is performed and the tension adjustment suture is pulled, when necessary, to achieve the desired continence. The mesh will lie in direct apposition to the urethra. The adjustment thread is then cut short and the vaginal incision is closed with an absorbable suture.
  Arms: SIS group

SUMMARY:
One in five women will undergo prolapse surgery in their lifetime, and there is a strong correlation between prolapse and urinary incontinence. Pelvic floor surgeons aspire to improve relevant quality of life outcomes for women with pelvic floor disorders while minimizing complications and unnecessary procedures. There has been an experience of disappointment and frustration when a patient returns following POP repair with new symptoms of Stress Urinary Incontinence (SUI) that she ranks as a greater disruption to her quality of life than her original vaginal bulge. While retropubic (RP) slings are considered to be the "gold-standard" referent for other slings with long-term outcomes data, they are associated with the highest risks of intra- and post-operative complications including bladder injury, bleeding, and post-operative voiding dysfunction. Single-incision slings (SIS) are the latest iteration in sling development that build upon the benefits of slings but avoid passage through the muscles of the inner thigh. The hypothesis for this study is that single-incision slings (Altis) are non-inferior to Retropubic mid-urethral slings when placed at the time of native tissue vaginal repair.

DETAILED DESCRIPTION:
Pelvic floor surgeons aspire to improve relevant quality of life outcomes for women with pelvic floor disorders while minimizing complications and unnecessary procedures. Efficacy and risk always compete for equilibrium. Level I evidence has demonstrated a positive efficacy benefit of a concomitant synthetic mid-urethral sling in women with, and without, pre-operative symptoms of SUI who are undergoing POP repair. Concomitant sling placement has been shown to reduce the risk of de novo or persistent SUI from 50% to 23%. The combination of surgical treatment of POP and SUI at the same time, however, increases the risk of incomplete bladder emptying. While retropubic (RP) slings are considered to be the "gold-standard" referent for other slings with long-term outcomes data, they are associated with the highest risks of intra- and post-operative complications including bladder injury, bleeding, and post-operative voiding dysfunction. Single-incision slings (SIS) are the latest iteration in sling development that build upon the benefits of slings but avoid passage through the muscles of the inner thigh. As the combination of POP and sling surgery increases the risk of voiding dysfunction, and rates of incomplete bladder emptying appear significantly lower for SIS than RP slings, the study team hypothesizes that the use of the Single-incision Mid-Urethral Sling SIS will be non-inferior to RP slings in efficacy and superior in irritative voiding symptoms/voiding dysfunction at one year after combined surgery.

ELIGIBILITY:
Inclusion Criteria:

* At least 21 years of age
* Women being considered for a native tissue vaginal repair in any vaginal compartment or colpocleisis
* POP ≥ stage II of any vaginal compartment, according to the pelvic organ prolapse quantification (POP-Q) system
* Vaginal bulge symptoms
* Positive standardized cough stress test on clinical examination, or on urodynamic testing
* Surgical plan that includes a native tissue vaginal repair including colpocleisis for symptomatic POP in any compartment
* Understanding and acceptance of the need to return for all scheduled follow-up visits
* English speaking and able to give informed consent
* Willing and able to complete all study questionnaires

Exclusion Criteria:

* Prior surgery for stress urinary incontinence
* Status post reconstructive pelvic surgery with transvaginal mesh kits or sacrocolpopexy with synthetic mesh for prolapse
* Any serious disease, or chronic condition, that could interfere with the study compliance
* Unwilling to have a synthetic sling
* Inability to give informed consent
* Pregnancy or planning pregnancy in the first postoperative year
* Untreated urinary tract infection (may be included after resolution)
* Poorly-controlled diabetes mellitus (HgbA1c > 9 within 3 months of surgery date)
* Prior pelvic radiation
* Incarcerated
* Neurogenic bladder/ pre-operative self-catheterization
* Elevated post-void residual (>150 ml) that does not resolve with prolapse reduction testing (pessary, prolapse reduced uroflow or micturition study)
* Prior augmented (synthetic mesh, autologous graft, xenograft, allograft) prolapse repair
* Planned concomitant bowel related surgery including sphincteroplasty and perineal rectal prolapse surgery, rectovaginal fistula repair, hemorrhoidectomy.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2018-12-12 (Actual); Primary Completion 2024-01-02 (Actual); Study Completion 2024-01-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Matthews, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (6):
- United States (6):
  - MedStar Health/National Center for Advance Pelvic Surgery, Washington D.C., District of Columbia
  - Northwestern Medical Group, Chicago, Illinois
  - Northwell Health, Manhasset, New York
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Women & Infants Hospital of Rhode Island, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mezes CM, Russell GB, Gutman RE, Iglesia C, Rardin C, Kenton K, Collins S, Matthews CA. Effect of Vaginal Prolapse Repair and Midurethral Sling on Urgency Incontinence Symptoms. Urogynecology (Phila). 2025 Mar 1;31(3):250-257. doi: 10.1097/SPV.0000000000001620. Epub 2024 Dec 13. PMID 39689213
- [Derived] Matthews CA, Rardin CR, Sokol A, Iglesia C, Collins S, Ferrando C, Winkler H, Kenton K, Geynisman-Tan J, Gutman RE. A randomized trial of retropubic vs single-incision sling among patients undergoing vaginal prolapse repair. Am J Obstet Gynecol. 2024 Aug;231(2):261.e1-261.e10. doi: 10.1016/j.ajog.2024.04.036. Epub 2024 May 3. PMID 38705225
- [Derived] Carter E, Johnson EE, Still M, Al-Assaf AS, Bryant A, Aluko P, Jeffery ST, Nambiar A. Single-incision sling operations for urinary incontinence in women. Cochrane Database Syst Rev. 2023 Oct 27;10(10):CD008709. doi: 10.1002/14651858.CD008709.pub4. PMID 37888839

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Total 280 patients signed the Informed Consent. Out of enrolled 280 patients, 3 withdrawn as screen failed, 21 dropped out before randomization, and 1 did not receive the treatment as per randomization. Hence enrolled number is larger than the randomized.
Period: Overall Study
Arm/Group | RP Sling Group | SIS Group
Started | 129 | 126
Completed | 122 | 118
Not Completed | 7 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RP Sling Group | SIS Group | Total
Number analyzed (Participants) | 129 | 126 | 255
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.5 (0) | 67.8 (0) | 67 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 129 | 126 | 255
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 4 | 10
  Not Hispanic or Latino | 123 | 121 | 244
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 11 | 24
  White | 112 | 111 | 223
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Subjectively Bothersome Stress Incontinence
Description: Dichotomous outcome (Yes/No), measured by a positive response of > 1 to Question 17 on Pelvic Floor Distress Inventory short form-20 (PFDI-20). Response scale from 0 to 4. Symptoms Not Present = NO 0 = not present Symptoms Present = YES, scale of bother: 1 = not at all, 2 = somewhat, 3 = moderately, 4 = quite a bit
Time Frame: 12 months post-operatively
Measure: Count of Participants; unit: Participants
Arm/Group | RP Sling Group | SIS Group
Number analyzed (Participants) | 129 | 126
Participants | 129 | 126

2. Primary Outcome: Count of Participants Needing Retreatment for Stress Incontinence
Description: This includes pelvic floor physical therapy; incontinence pessary; urethral bulking injection; repeat incontinence surgery.
Time Frame: 12 months post-operatively
Measure: Count of Participants; unit: Participants
Arm/Group | RP Sling Group | SIS Group
Number analyzed (Participants) | 122 | 118
Participants | 3 | 5

3. Primary Outcome: Count of Participants With De Novo or Worsening Urge Incontinence Symptoms
Description: Dichotomous outcome (Yes/No), measured by a worsening change in response to Question 16 on PFDI-20 with at least somewhat bothersome symptoms. Response scale from 0 to 4. Symptoms Not Present = NO 0 = not present Symptoms Present = YES, scale of bother: 1 = not at all, 2 = somewhat, 3 = moderately, 4 = quite a bit
Time Frame: 12 months post-operatively
Measure: Count of Participants; unit: Participants
Arm/Group | RP Sling Group | SIS Group
Number analyzed (Participants) | 109 | 103
Participants | 3 | 3

4. Primary Outcome: Count of Participants Requiring Bladder Drainage
Description: Beyond 2 weeks post-operatively with PVR > 150 ml OR > 1/3 total voided volume up to 12 Month post-operatively..
Time Frame: 12 Month post-operatively
Measure: Count of Participants; unit: Participants
Arm/Group | RP Sling Group | SIS Group
Number analyzed (Participants) | 109 | 103
Participants | 0 | 0

5. Primary Outcome: Count of Participants Needing Surgical Intervention for Urinary Retention
Description: Sling lysis or revision at any time point post-operatively up to 12 Month post-operatively.
Time Frame: 12 Month post-operatively
Measure: Number; unit: participants
Arm/Group | RP Sling Group | SIS Group
Number analyzed (Participants) | 109 | 103
participants | 3 | 4

6. Secondary Outcome: Number of Participants With Adverse Events
Description: Reporting of adverse events intra- and post-operatively and include adverse events as measured by the Dindo classification system.
Time Frame: 12 months post-operatively
Measure: Number; unit: Participants with Adverse Events
Arm/Group | RP Sling Group | SIS Group
Number analyzed (Participants) | 109 | 103
Participants with Adverse Events | 47 | 53

7. Secondary Outcome: Surgeon Satisfaction Scores
Description: Surgeon satisfaction with the sling will be assessed with a 10-point Likert Scale. The scale has a score range of 0-10, with 0=no satisfaction 10=extremely satisfied.
Time Frame: post-operatively up to 12 months
Measure: Mean (Full Range); unit: Score on a Scale
Arm/Group | RP Sling Group | SIS Group
Number analyzed (Participants) | 129 | 126
Score on a Scale | 9 [8 to 10] | 8 [7 to 10]

ADVERSE EVENTS:
Time Frame: 1 year
Description: Protocol defined urogynecologic adverse events collected.
Arm/Group | RP Sling Group | SIS Group
All-Cause Mortality (participants affected / at risk) | 0/129 | 0/126
Serious Adverse Events (participants affected / at risk) | 7/129 | 6/126
Other Adverse Events (participants affected / at risk) | 40/129 | 47/126
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RP Sling Group (N=129) | SIS Group (N=126)
Voiding Dysfunction (Surgical and medical procedures) | 2 (2) | 2 (2) — Voiding Dysfunction led to sling lysis
Urosepsis (Surgical and medical procedures) | 1 (1) | 0 (0)
Pelvic Abscess (Infections and infestations) | 1 (1) | 0 (0)
Pelvic Hematoma (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Recurrent Prolapse (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Pelvic Pain (Surgical and medical procedures) | 0 (0) | 1 (1)
Death (Surgical and medical procedures) | 0 (0) | 0 (0)
Urinary Retention (Surgical and medical procedures) | 2 (2) | 2 (2) — Urinary Retention leading to Sling Lysis
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RP Sling Group (N=129) | SIS Group (N=126)
Bleeding (Surgical and medical procedures) | 2 (2) | 5 (5)
Hematoma (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Infection (Infections and infestations) | 5 (5) | 1 (1) — Vaginal // Pelvic Abscess
Mesh Exposure (Surgical and medical procedures) | 0 (0) | 1 (1)
Recurrent POP (Congenital, familial and genetic disorders) | 1 (1) | 2 (2) — POP = Pelvic Organ Prolapse
Readmission for Complications (Surgical and medical procedures) | 2 (2) | 2 (2)
Outpatient Surgical Intervention (Surgical and medical procedures) | 3 (3) | 4 (4)
Urinary Tract Infection (Infections and infestations) | 15 (15) | 25 (25)
Urgency "De Novo" (Renal and urinary disorders) | 3 (3) | 3 (3)
Voiding Dysfunction (Renal and urinary disorders) | 5 (5) | 4 (4)
Leg Pain (Surgical and medical procedures) | 1 (1) | 0 (0)
Bowel Injury (Surgical and medical procedures) | 0 (0) | 0 (0)
Bowel Obstruction (Surgical and medical procedures) | 0 (0) | 0 (0)
Fistula (Surgical and medical procedures) | 0 (0) | 0 (0)
Intestinal Injury (Surgical and medical procedures) | 0 (0) | 0 (0)
Mesh Erosion (Surgical and medical procedures) | 0 (0) | 0 (0)
Nerve Injury (Surgical and medical procedures) | 0 (0) | 0 (0)
Venous Thromboembolism (Surgical and medical procedures) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-01-10): https://cdn.clinicaltrials.gov/large-docs/14/NCT03520114/Prot_001.pdf
  • Informed Consent Form (2022-03-16): https://cdn.clinicaltrials.gov/large-docs/14/NCT03520114/ICF_000.pdf